CLINICAL TRIAL: NCT06484517
Title: Is HugeMed Video Laryngoscope Superior to McGrath in Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Gamze Tanırgan Çabaklı, Dr., Marmara University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Device Feasibility
Other Study IDs: 09.2021.961
Record Dates: First submitted 2024-06-16; First posted 2024-07-03 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2024-07

CONDITIONS: Difficult Intubation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The group of patients (Group M, n=20) was intubated with the McGrath videolaryngoscope. (Active Comparator): Before intubation, Cormack-Lehane score and percentage of glottis opening (POGO) score were recorded by applying direct and indirect laryngoscopy with the Macgreth videolaryngoscope. All tracheal intubations were performed by the same expert with over 10 years of experience in pediatric anesthesia.
  Interventions: Device: Hugemed Videolaryngoscope
- For the group (Group H, n=20), the Hugemed videolaryngoscope was used. (Experimental): Patients were intubated using one of the appropriate blades numbered 1, 2, or 3 based on their height, weight, and age. After the induction of general anesthesia, patients underwent direct and indirect laryngoscopy with videolaryngoscopes. The Modified Cormack-Lehane score and Percentage of Glottic Opening (POGO) score were recorded, and orotracheal intubation was performed. Number of attempts, need for cricoid pressure, optimization maneuvers, success rate, and hemodynamic parameters of both groups were recorded.
  Interventions: Device: Hugemed Videolaryngoscope

INTERVENTIONS:
Device: Hugemed Videolaryngoscope — After general anesthesia induction, the first group of patients (Group M, n=20) was intubated with the McGrath videolaryngoscope. For the second group (Group H, n=20), the Hugemed videolaryngoscope was used. Patients were intubated using one of the appropriate blades numbered 1, 2, or 3 based on their height, weight, and age.
  Other Names: Mc Grath Videolaryngoscope

SUMMARY:
Videolaryngoscopes improve laryngeal visualization in children under 3 years. In this study we aimed to compare Hugemed and McGrath videolaryngoscopes regarding their Cormach-Lehane (CL) and percentage of glottic opening (POGO) scores. Furthermore, tracheal intubation success rates, need for cricoid pressure and optimization maneuvers, and hemodynamic changes are compared.

ELIGIBILITY:
Inclusion Criteria:

total of 40 elective surgical patients under the age of 3, classified as ASA 1-3 risk group, who underwent general anesthesia with no anticipated difficult airway.

Exclusion Criteria:

Patients who could not obtain parental consent, those classified as ASA 4 and above, individuals with serious cardiac and respiratory problems, and patients anticipated to have a difficult airway were not included in the study.

Ages: 6 Months to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Success of intubation | Procedure (At the time of the intubation of the patient.)
  Number of attempts of the intubation.

SECONDARY OUTCOMES:
Percentage of glottis opening (POGO) | Procedure (At the time of the intubation of the patient.)
  The primary aim of this study was to compare the percentage of glottis opening (POGO, 0-100%) scores in direct and indirect laryngoscopy performed with HugeMed and McGrath video laryngoscopes in pediatric patients.
Need for optimization maneuvers | Procedure (At the time of the intubation of the patient.)
  Whether there are any optimization maneuvers by an assistant.
Degree of hemodynamic changes | Procedure (At the time of the intubation of the patient.)
  Whether there are any acute changes in the patient heart rate during the intubation.
blood pressure | Procedure (At the time of the intubation of the patient.)
  Whether there are any acute changes in the patient blood pressure during the intubation.
Success of intubation | Procedure (At the time of the intubation of the patient.)
  Number of attempts of the intubation.

CONTACTS AND LOCATIONS:
Overall Officials: Gamze Çabaklı, Principal Investigator — Marmara University Department of Anesthesiology and Reanimation
Locations (1):
- Marmara University Pendik Research and Training Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cabakli GT, Saracoglu KT, Abdullayev R, Guclu E, Ratajczyk P, Saracoglu A. A Comparison of McGrath Mac and HugeMed Video Laryngoscopes in Pediatric Patients Under 3 Years Old-A Prospective Randomized Trial. Healthcare (Basel). 2025 Apr 7;13(7):842. doi: 10.3390/healthcare13070842. PMID 40218139